CLINICAL TRIAL: NCT07012707
Title: Rationale and Trial Design of PFB-03 Study: Diagnostic Performance and Clinical Application of 18F-FAPI-PET/CT for Detecting Axillary Lymph Node Metastasis in Breast Cancer Patients After Neoadjuvant Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, ZHOU Yidong, Chief of Dept. Breast Surgery, Peking Union Medical College Hospital
Other Study IDs: PUMCH-PFB03
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Double positive: If clinical exam and 18F-FAPI PET/CT are positive for ALN involvement both before and after NAT, the patient proceeds directly to ALND as per standard guidelines.
- Single Positive: If clinically/pathologically node-positive (c/pN1) pre-NAT but becomes clinically and 18F-FAPI PET/CT negative post-NAT, the patient undergoes ALND as per standard guidelines. However, within this ALND procedure, sentinel lymph nodes (SLNs) will be identified and sent separately for pathological analysis to assess the FNR of FAPI-PET guided SLNB evaluation in this specific scenario, without additional trauma or cost to the patient.
- Double Negative: Includes two subgroups: (a) Patients who were clinically/pathologically node-negative pre-NAT and remain clinically and 18F-FAPI PET/CT negative post-NAT. (b) Patients who were clinically node-negative pre- and post-NAT, but 18F-FAPI-PET/CT becomes positive post-NAT. Within Cohort 3, management depends on patient preference: either proceed directly to ALND or undergo SLNB first (using dual tracer). If SLNB is positive, completion ALND follows; if negative, ALND is omitted. Dual tracer methods include methylene blue, contrast-enhanced ultrasound, or radionuclide imaging.

SUMMARY:
Axillary lymph node (ALN) status is a crucial prognostic factor in breast cancer. Accurate, non-invasive methods for evaluating axillary lymph node metastasis after neoadjuvant therapy (NAT) are needed to optimize surgical decisions and minimize patient morbidity. Fibroblast Activation Protein Inhibitor (FAPI) PET/CT targets cancer-associated fibroblasts and may improve diagnostic accuracy. This study aims to assess the diagnostic performance and clinical utility of 18F-FAPI PET/CT in detecting ALN metastasis after NAT in breast cancer patients. This prospective, single-center study will enroll breast cancer patients with cT1-4N0-1M0 stage before NAT, who will undergo pre-surgical 18F-FAPI PET/CT followed by sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND) guided by protocol stratification based on FAPI PET/CT and clinical findings. The primary endpoint is the diagnostic accuracy of 18F-FAPI PET/CT for ALN metastasis versus pathology. Secondary endpoints include false-negative rates (FNR) of SLNB, lymphedema rates, and long-term outcomes such as local recurrence and survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent
* Female at 18-80 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* With anticipated survival of at least 36 months
* Pathologically confirmed invasive breast cancer with clinical stage of T1-4N0-1M0
* Received standard NAT for BC (including either neoadjuvant chemotherapy or neoadjuvant targeted therapy, or a combination)
* Have willingness to take the 18F-FAPI PET/CT imaging
* With adequate organ function (neutrophil count ≥ 1.5 × 10⁹/L; platelet count ≥ 90 × 10⁹/L; hemoglobin ≥ 90 g/L; total bilirubin ≤ 1.5 × upper limit of normal [ULN]; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; blood urea nitrogen (BUN) and serum creatinine (Cr) ≤ 1.5 × ULN; international normalized ratio (INR) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN).

Exclusion Criteria:

* Evidence of distant metastatic disease (M1)
* Pregnant or lactating women
* Failure to complete the planned NAT
* Prior surgical intervention in the ipsilateral axilla
* Diagnosis of any other malignancy within the past 5 years (exceptions: adequately treated non-melanoma skin cancer, cervical carcinoma in situ, papillary thyroid cancer)
* Known hypersensitivity to the FAPI tracer or any excipients
* With any serious uncontrolled medical condition that would make the patient unsuitable for surgery or PET/CT (e.g. unstable cardiac disease, severe claustrophobia unresponsive to anxiolytics, renal failure preventing CT contrast if needed)
* Failure to lie still for imaging (about 20-30 minutes) or adhere to follow-up due to psychiatric, cognitive, or social reasons.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed as a single-center, prospective observational diagnostic accuracy trial. It will be conducted at the Department of Breast Sugery and Nuclear Medicine of PUMCH, Beijing, China, between June 2025 and May 2027. The study population consists of stage cT1-4N0-1M0 breast cancer patients with who received NAT (Fig. 1). After completion of NAT, surgical approach (ALND/SLNB) is guided by protocol stratification based on 18F-FAPI PET/CT and clinical findings. There is no randomization in this study, and all enrolled patients will undergo the index test and the reference standard surgical evaluation.
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of 18F-FAPI PET/CT for detecting residual axillary lymph node metastases after NAT | Through study completion, an average of 3 years.
  The primary endpoint of the study is the diagnostic accuracy of 18F-FAPI PET/CT for detecting residual axillary lymph node metastases after NAT, on a patient-level analysis. This will be assessed by calculating:
  i)Sensitivity: proportion of patients with pathologically proven residual nodal metastasis who had a positive 18F-FAPI PET/CT (true positive rate).
  ii)Specificity: proportion of patients with no residual nodal metastasis (pathologic nodal pCR) who had a negative PET/CT (true negative rate).
  iii)Positive predictive value (PPV): probability that a PET-positive patient truly has nodal disease on pathology.
  iv)Negative predictive value (NPV): probability that a PET-negative patient is truly node-negative on pathology.
  v)Overall accuracy: proportion of all patients correctly classified by PET (true positives + true negatives divided by total).

IPD SHARING:
Plan to Share IPD: No